CLINICAL TRIAL: NCT00457899
Title: RAPID-An Open-Label Randomized, Multicenter Phase IIIb Study to Evaluate the Efficacy and Tolerability of Quetiapine IR (Immediate Release), Over 14 Days, in Acute Schizophrenia/Schizoaffective Disorder (Rapid Versus Conventional Titration)
Brief Title: Rapid Versus Conventional Titration of Quetiapine in Schizophrenia/Schizoaffective Disorder
Acronym: RAPID
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to poor recruitment
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00003
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Schizophrenia; Schizoaffective Disorders; Psychotic Disorders
Keywords: schizophrenia; schizoaffective disorder; quetiapine; seroquel; titration
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine IR (Immediate Release) — oral
  Other Names: Seroquel

SUMMARY:
The purpose of this study is to determine whether increasing the amount (dose) of quetiapine IR (immediate release formulation) more rapidly than conventional dose increases, improves the control of symptoms as measured by the Positive and Negative Syndrome Scale (PANSS) - a psychiatric assessment scale that measures both positive and negative symptoms - in patients with acute schizophrenia or schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 to 65 years, who require treatment for an acute episode of schizophrenia/schizoaffective disorder as judged by their doctor

Exclusion Criteria:

* Significant and unstable conditions of hear, circulation, blood, liver, kidney; malignancies (cancer); diabetes (mellitus); history of fits or fainting. Resistance to antipsychotic medication. Current alcohol/drug abuse. Pregnant/breast feeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2007-07; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable of this study is change from baseline in total PANSS score | at Day 7

SECONDARY OUTCOMES:
Change from baseline in total PANSS scores | on day 5 and 14
change from baseline in CGI-S and absolute CGI-I | on days 5, 7 and 14
frequency and severity of adverse events; change in vital signs. | assessed at each visit
change from baseline in subscale PANSS and PANSS-EC scores | on days 5, 7 and 14

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca UK Medical Director, MD, Study Director — AstraZeneca UK; Professor Gary Sullivan, MD, Principal Investigator — St Tydfil's Hospital
Locations (12):
- United Kingdom (12):
  - Research Site, Brentwood, Essex
  - Research Site, Harrow, Middlesex
  - Research Site, Surbiton, Surrey
  - Research Site, Birmingham
  - Research Site, Bognor Regis
  - Research Site, Bury St Edmunds
  - Research Site, Coventry
  - Research Site, Crewe
  - Research Site, Darlington
  - Research Site, London
  - Research Site, Sandbach
  - Research Site, Warrington